CLINICAL TRIAL: NCT04457934
Title: Effectiveness of PLENVU in the General Screening Population and Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Prof. Helmut Neumann, Head of Interdisciplinary Endoscopy, Johannes Gutenberg University Mainz
Other Study IDs: 001; 125 (Other Grant/Funding Number: Norgine)
Record Dates: First submitted 2020-06-15; First posted 2020-07-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: IBD; Healthy
Keywords: endoscopy; preparation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD patients: Patients with IBD will undergo preparation for Standard endoscopy with PLENVU, since it is considered to be less affecting for patients. IBD patients have to undergo endoscopy often and mostly suffer from non-efficient preparation.
  Patients will drink 1 Liter of Plenvu and 1 Liter of water or tea in preparation for endoscopy and will follow the Guidelines for preparation of endoscopy.
  The only Change from Standard care is that patients will receive Plenvu instead of Movicol.
  Interventions: Drug: Plenvu
- Screening patients: Screening patients will undergo Standard endoscopy to prevent colon Cancer. Patients will drink 1 Liter of Plenvu and 1 Liter of water or tea in preparation for endoscopy and nd will follow the Guidelines for preparation of endoscopy.
  The only Change from Standard care is that patients will receive Plenvu instead of Movicol.
  Interventions: Drug: Plenvu

INTERVENTIONS:
Drug: Plenvu — All patients in both Groups will drink will drink 1 Liter of Plenvu and 1 Liter of water or tea in preparation for endoscopy according to endoscopy guidelines

SUMMARY:
Patients presenting for endoscopic surveillance of IBD or colorectal screening colonoscopy at one of the participating centers will be asked to participate in the present study after careful evaluation of inclusion and exclusion criteria. The aim is that the final study population will comprise of 50% IBD patients and 50% colorectal cancer screening patients. Before inclusion, all patients have to sign the written informed consent. All participating patients will receive PLENVU, a well-known and approved bowel preparation agent. Bowel preparation is performed following the general recommendations of use. Following the bowel preparation, patients are asked if they have well tolerated the preparation, if they already had a colonoscopy in the past with another bowel preparation agent and if they would prefer PLENVU or another bowel preparation for their next endoscopy examination. Endoscopy is performed in standard way and effectiveness of the bowel preparation is specifically highlighted by the physician on the documentation report. Finally, data is analyzed regarding effectiveness of PLENVU for bowel preparation and patient satisfaction.

DETAILED DESCRIPTION:
PLENVU is effective for bowel preparation and the efficacy and safety of PLENVU has been investigated in randomized controlled trials in patients undergoing gut cleansing prior to colonoscopy. Data on the specific screening population and for patients suffering from IBD however is limited to date. The aim of the current study is to fill this gap and to provide data of the effectiveness of PLENVU for the specific patients groups in order to provide specific recommendations for an adequate bowel preparation in those groups.

In general, bowel-preparation in IBD patients is often more challenging. This might be due to the chronic disease burden but also according to compliance factors of individual patients. Of note, an adequate bowel-preparation is of paramount importance in IBD in order to detect subtle neoplasia and to perform chromoendoscopy, which is still recommended by the updated ESGE guideline.

It is anticipated, that PLENVU will help IBD patients to achieve a better bowel preparation, thereby yielding in more effective screening colonoscopies and higher acceptance rates of patients for surveillance colonoscopies. In order to show that no significant differences are seen in the included IBD cohort compared to the general screening population (bias risk), the investigators aim to also include patients from the normal screening population.

ELIGIBILITY:
Inclusion Criteria:

* • Suspicion or history of IBD

  * Screening colonoscopy
  * Indication for colonoscopy
  * Age 18-75 years
  * Written informed consent

Exclusion Criteria:

* • Pregnancy or lactating

  * Lower gastrointestinal bleeding with hemodynamic instability
  * Bowel obstruction
  * ASA >3
  * Not sufficiently corrected anticoagulation disorders
  * Plenvu must not be taken:

    * if you are allergic (hypersensitive) to the active ingredients or any of the other ingredients of this medicine;
    * if you have a blockage (obstruction) in the digestive tract.
    * if you have a breakthrough (perforation) in the wall of the digestive tract;
    * if you suffer from intestinal obstruction (Ileus);
    * if you suffer from a disturbance of gastric emptying (e.g. gastroparesis, gastric retention);
    * if you suffer from phenylketonuria. Phenylketonuria is a congenital metabolic disease in which phenylalanine cannot be processed by your body. Plenvu contains aspartame as a source of phenylalanine;
    * if you suffer from glucose-6-phosphate dehydrogenase deficiency;
    * if you suffer from acute colon enlargement (toxic megacolon).
  * Warnings and precautions

    o You should tell your doctor about the following circumstances before taking Plenvu:
  * if you have heart problems and/or arrhythmias;
  * if you have kidney problems and/or suffer from dehydration;
  * if you have stomach or intestinal problems, including intestinal inflammation;
  * if you have difficulty or discomfort when swallowing liquids;
  * if you have high or low levels of electrolyte (e.g. sodium, potassium);
  * if you have other diseases (e.g. convulsions).
  * Pregnancy and lactation o There are no data on the use of Plenvu during pregnancy or lactation and is therefore not recommended.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Screening colonoscopy; IBD; age group 18-75 years
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Standard (BBPS) | 1 week
  Bowel preparation according to international Standard (1 is bad, 9 is good), how many BBPs with 9 can be achieved?
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 day
  How good will patients tolerate endoscopy and preparation
Number of patients with adverse events | up to 1 week
  What Kind of adverse Events can happen during this study

SECONDARY OUTCOMES:
Number of patients who are willing to accept repeated examination (surveillance); | up to 1 month
  How many patients will come back for another endoscopy
Adenoma and Polyp Detection Rate (ADR and PDR) | 1 day
  How many adenomas and polyps are detected during endoscopy
cecal intubation rate | 1 day
  how many endoscopies will reach the ceacum
procedure time | 3 hours
  how Long will endoscopy take

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, Prof. Dr., Principal Investigator — University Medical Center Mainz
Locations (3):
- Germany (3):
  - Dr. Helmut Neumann, Bad Salzuflen, Northrine-Westfalia
  - Dr. Horst Hohn, Koblenz, Rhenanie-Palatinate
  - University Hospital Mainz, Mainz

IPD SHARING:
Plan to Share IPD: Yes
* Preliminary data 2020 for: DDW 2021 (Deadline Dec. 1st), preliminary data will be available for Norgine for DGVS (Germany) and APDW (Malaysia).
  * Final data: Submission 2021 for DDW, ESGE Days, UEGW, DGVS, APDW
  * Final manuscript: Am J Gastro -> Journal Crohn's Colitis -> Endoscopy -> Gastrointest Endos
Supporting Information: Study Protocol, ICF
Time Frame: January 2021-December 2021
Access Criteria: Abstracts and publications